CLINICAL TRIAL: NCT01490723
Title: Dose-Intense Yttrium-90 Ibritumomab Tiuxetan (Zevalin)-Containing Non-Myeloablative Conditioning for Allogeneic Stem Cell Transplantation in B-cell Malignancies
Brief Title: Zevalin-Containing Nonmyeloablative Conditioning for Stem Cell Transplantation (SCT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0393; NCI-2016-00250 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-12-09; First posted 2011-12-13 (Estimated); Results first posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Leukemia; Lymphoma
Keywords: Leukemia; Chronic lymphocytic leukemia; Lymphoma; CD20+ lymphoid malignancies; Diffuse large B-cell lymphoma; Allogeneic transplantation; Rituximab; Rituxan; In ibritumomab; Y ibritumomab; Zevalin; Fludarabine Phosphate; Fludara; Bendamustine Hydrochloride; Bendamustine HCL; CEP-18083; SDX-105; Treanda; Stem Cell Transplantation; Planar Scintigraphy; Spect Scan; Single Photon Emission-Computed Tomography; CT Scan; Computed Tomography; G-CSF; Filgrastim; Neupogen; Thymoglobulin; ATG; Antithymocyte Globulin; Methotrexate; Mycophenolate; MMF; Mycophenolate Mofetil; CellCept; Tacrolimus; Prograf
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; ibritumomab tiuxetan; fludarabine; fludarabine phosphate; Bendamustine Hydrochloride; thymoglobulin; Antilymphocyte Serum; Tacrolimus; Methotrexate; Mycophenolic Acid; Granulocyte Colony-Stimulating Factor; Filgrastim; Stem Cell Transplantation; Transplantation, Homologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Yttrium-90 Ibritumomab + Chemo (Experimental): Day -22 and -14, Rituximab 250 mg/m2 preceding 111In Ibritumomab and (90Y) ibritumomab tiuxetan administration, respectively. Day -22, -21 to -16, Imaging, repeated 3-6 hours later (including Single Photon Emission-Computed Tomography/Computed Tomography (SPECT/CT) scan of the abdomen). Day -14, (90Y) ibritumomab tiuxetan administration. Day -5, -4 and -3, Fludarabine and Bendamustine following Stem Cell Transplant (SCT) and CT. Fludarabine 30 mg/m2 intravenously followed by Bendamustine 130 mg/m2 intravenously. All patients receive Graft Versus Host Disease (GvHD) prophylaxis, infections disease prophylaxis, growth factors, blood and platelet transfusion and other supportive treatment.
  Interventions: Drug: Rituximab; Drug: 111In Ibritumomab; Procedure: Planar Scintigraphy Imaging; Drug: 90Y IbritumomabTiuxetan; Drug: Fludarabine; Drug: Bendamustine; Drug: Thymoglobulin; Drug: Tacrolimus; Drug: Methotrexate; Drug: Mycophenolate; Drug: G-CSF; Procedure: Stem Cell Transplantation

INTERVENTIONS:
Drug: Rituximab — 250 mg/m2 by vein preceding 111In Ibritumomab and (90Y) ibritumomab tiuxetan administration, respectively on Days -22 and -14.
  Other Names: Rituxan
Drug: 111In Ibritumomab — (5.0 mCi +/- 10% of 111In) by vein immediately following the infusion of rituximab on Day -22.
  Other Names: Zevalin
Procedure: Planar Scintigraphy Imaging — Day -22, -21 to -16: Planar scintigraphy whole-body imaging started on Day -22 post 111In Ibritumomab infusion prior to voiding, and repeated 3-6 hours later (including Single Photon Emission-Computed Tomography/Computed Tomography (SPECT/CT) scan of the abdomen). Whole-body planar scintigraphy imaging will be repeated between 22-26 hours, then between 70-74 hours, and later between 142-146 hours post 111In Ibritumomab injection.
Drug: 90Y IbritumomabTiuxetan — Calculated to deliver not below 10 Gy to normal organs (liver, lungs, kidneys) by vein post rituximab on Day -14.
  Other Names: Zevalin
Drug: Fludarabine — 30 mg/m2 intravenously on Days -5, -4, and -3.
  Other Names: Fludarabine Phosphate; Fludara
Drug: Bendamustine — 130 mg/m2 intravenously on D-5, -4 and -3.
  Other Names: Bendamustine Hydrochoride; Bendamustine HCL; CEP-18083; SDX-105; Treanda
Drug: Thymoglobulin — 1 mg/kg (based on actual body weight) on Days -2 and -1 will be administrated to patients receiving a cord blood (CB) and a matched unrelated donor (MUD).
  Other Names: ATG; Antithymocyte Globulin
Drug: Tacrolimus — Starting dose of 0.015 mg/kg (ideal body weight) as a 24 hour continuous infusion daily adjusted to achieve a therapeutic level of 5-15 ng/ml. Tacrolimus is changed to oral dosing when tolerated and can be tapered off after day +90 if no Graft versus Host Disease (GVHD) is present.
  For patients receiving cord blood (CB) graft, the Graft versus Host Disease (GvHD) prophylaxis will be with Tacrolimus. Tacrolimus will start on D-2 administrated at starting dose 0.03 mg/kg or 0.015 mg/kg (ideal body weight) by vein starting on D -2 and will be tapered around Day +180 if no GvHD is present.
  Other Names: Prograf
Drug: Methotrexate — 5 mg/m2 by vein on Day +1, +3 and +6. Patients receiving an unrelated graft will also be given methotrexate on Day +11 after the transplant.
Drug: Mycophenolate — 15 mg/kg (actual body weight with a maximum dose of 1 gram twice daily) by vein or by mouth administered from Days -3 to +45 and then tapered to end by day 100 if there is no Graft versus Host Disease (GVHD).
  Other Names: MMF; Mycophenolate Mofetil; CellCept
Drug: G-CSF — 5 mcg/kg/day subcutaneously beginning Day +7 for patients receiving related and matched unrelated donor (MUD) grafts and on Day 0 for patients receiving a cord blood (CB). G-CSF will continue until the absolute neutrophil count (ANC) is > 500 * 10/L for 3 consecutive days.
  Other Names: Filgrastim; Neupogen
Procedure: Stem Cell Transplantation — Stem Cell Transplantation on Day 0
  Other Names: Allogeneic transplantation

SUMMARY:
The goal of this clinical research study is to learn if adding Zevalin (ibritumomab tiuxetan) to low-intensity chemotherapy (the combination of rituximab, bendamustine, and fludarabine), followed by an allogeneic stem cell transplant, can help to control lymphoma. The safety of this combination will also be studied.

Two (2) forms of ibritumomab tiuxetan will be used in this study. 90Y-ibritumomab tiuxetan is designed to attach to lymphoma cells and destroy the cells using a radioactive particle that is attached to it. 111In-ibritumomab tiuxetan is like 90Y- ibritumomab tiuxetan, but the radioactive particle that is attached to it does not kill lymphoma cells. The radioactive particle makes the drug able to be seen inside your body. It is being used in this study to predict how fast the study drug will travel in the body and how long the drug stays in the body.

Rituximab is designed to attach to lymphoma cells, which may cause them to die.

Bendamustine is designed to damage and destroy the DNA (genetic material) of cancer cells.

Fludarabine is designed to make cancer cells less able to repair damaged DNA. This may increase the likelihood of the cells dying.

DETAILED DESCRIPTION:
Study Drug Administration and Procedures:

The chemotherapy, some of the other drugs in this study, and the stem cell transplant will be given by vein through your central venous catheter (CVC). A central venous catheter is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia and will remain in your body during treatment. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form. Blood samples will also be drawn through the CVC.

On Days -22 (22 days before you receive the stem cell transplant), you will receive rituximab by vein over 3-4 hours. You will then receive 111In-ibritumomab tiuxetan by vein over 30 minutes.

From Day -22 through Day -16, you will have scans called whole-body planar scintigraphy imaging. In these scans, a special camera will capture 2-dimensional images of the whole body to see where the radioactive 111In- ibritumomab tiuxetan that was injected on Day -22 has spread. No additional radiation will be used in this scan. Scintigraphy will be performed right after the injection, then 3-6 hours after the injection, then 24, 72, and 144 hours (+/- 2 hours) after the injection.

After the last scintigraphy imaging scan, the scans will be reviewed to learn how much radiation has traveled to different organs and to decide how much 90Y- ibritumomab should be used.

On Day-14, you will receive rituximab by vein over 3-4 hours. You will then receive the calculated dose of 90Y-ibritumomab tiuxetan by vein over 30 minutes.

On Days -5, -4, and -3, you will receive fludarabine and bendamustine by vein over 1 hour each day.

On Days -3 through Day 100, if your stem cells are from cord blood, you will receive mycophenolate mofetil (MMF) by vein or by mouth. MMF is designed to block the donor cells from growing and spreading in a way that could cause graft versus host disease (GVHD -- a condition in which transplanted tissue attacks the recipient's body).

Starting on Day -2, if your stem cells are from a related or matched unrelated donor, you will receive tacrolimus by vein as a continuous (nonstop) infusion until you are able to take it by mouth to help prevent GVHD. You will then take tacrolimus by mouth 2 times a day for about 3 months. After that, your tacrolimus dose may be lowered if you do not have GVHD. Your doctor will discuss this with you.

On Days -2 and -1, if your stems cells are from a matched unrelated donor or from cord blood, you will receive thymoglobulin (ATG) by vein over about 4 hours. ATG is designed to weaken your immune system to reduce the risk of rejecting of the transplant.

On Day 0, you will receive the blood stem cells by vein over about 30-45 minutes. Blood (less than 1 teaspoon) will also be drawn to measure how much (if any) radiation from the 90Y- ibritumomab tiuxetan is left in the blood.

Starting on Day 0, if your stem cells are from cord blood, you will receive filgrastim (G-CSF) through a needle under the skin 1 time a day every day until your white blood count begins to recover. G-CSF is designed to help cells in the bone marrow to divide, which helps raise white blood cells counts more quickly, lower fever, and decrease the risk of infection.

On Days 1, 3, and 6, if your stem cells are from a related or matched unrelated donor, you will receive methotrexate over 30 minutes each day by vein to help prevent GVHD. Patients receiving a matched unrelated donor will also be given methotrexate on Day 11 after the transplant.

Starting on Day 7, if your stem cells are from a related or matched unrelated donor, you will receive G-CSF through a needle under the skin 1 time a day every day until your white blood count begins to recover.

When your doctor thinks they are needed, you will also receive antibiotics and antifungal drugs to help prevent and/or treat infections. Your doctor will tell you more about how these drugs are given and possible side effects.

You will be in the hospital for about 3-4 weeks after you receive the stem cell transplant. During this time, the following tests and procedures will be performed at any point that your doctor thinks they are needed:

* You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate).
* You will be asked about how you are feeling and about any side effects you may be having.
* Blood (about 4-6 teaspoons) will be collected for routine tests, to check your kidney and liver function, and to learn if and how well the transplant is working.

The following may also be performed if at any point the doctor thinks they are needed:

* You may have imaging scans to check the status of the disease and/or to check for possible infections.
* You may have a bone marrow biopsy to check the status of the disease. To collect a bone marrow biopsy, an area of the hip or other site is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a needle.
* You may have transfusions of blood and/or platelets.

You must stay in the Houston area for about 100 days after the stem cell transplant.

Long-Term Follow-Up:

About 3, 6, and 12 months after the stem cell transplant:

* Blood (about 6 teaspoons) will be collected for routine tests, to check kidney and liver function, and to see how well the transplant has taken.
* You will have CT and PET scans to check the status of the disease.
* You will have a bone marrow biopsy/aspirate to check the status of the disease.

About 2 and 3 years after the stem cell transplant, you will receive a phone call that will take less than 10 minutes to learn how you are doing.

Length of Study:

You will be on study for up to about 3 years. You may be taken off study early if the disease gets worse, if you have any intolerable side effects, of if you are unable to follow study directions.

You should talk to the study doctor if you want to leave the study early. If you are taken off study early, you still may need to return for routine post-transplant follow-up visits, if your transplant doctor decides it is needed. It may be life-threatening to leave the study after you have begun to receive the study drugs but before you receive the stem cells.

This is an investigational study. Ibritumomab tiuxetan, rituximab, bendamustine, and fludarabine are FDA approved and commercially available for the treatment of lymphoma. The dose of ibritumomab tiuxetan in this study is designed to be higher than the FDA approved dose. The use of ibritumomab tiuxetan and bendamustine in combination with the other study drugs and a stem cell transplant for the treatment of lymphoma is investigational.

Up to 20 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 70 years of age.
2. Patients with the following CD20+ lymphoid malignancies who are eligible for allogeneic transplantation: a. Relapsed or refractory follicular lymphoma; b. Relapsed or refractory or high risk mantle cell lymphoma (hi ki67; blastic); c. Recurrent or refractory marginal zone; d. Recurrent or refractory CLL/small lymphocytic lymphoma; e. Double-hit lymphoma; f. Diffuse large B cell lymphoma; g. Richter's patients; or h. Refractory or recurrent Burkitts.
3. Patients who meet criterion #2 or have any of the following are eligible: a. Less than PR to salvage chemotherapy; b. Kinetic failure; c. Having received more than 3 lines of therapy; d. Failure to mobilize autologous stem cell; e. 10% or more marrow involvement; f. 6 months post autologous stem cell transplant.
4. Patients must have a fully-matched related donor or a matched unrelated donor identified. Double cord (at least 4/6 matched) can be used if no adult matched donor is available.
5. Performance score of at least 80% by Karnofsky or 0 to 2 ECOG.
6. Left ventricular EF >/= 45% with no uncontrolled arrythmias or symptomatic heart disease.
7. FEV1, FVC >/= 60% and corrected DLCO >/= 60%.
8. Serum creatinine </=1.6 mg/dL. Serum bilirubin < 2 mg/dL (unless due to Gilbert's Syndrome).
9. SGPT < 2 X upper limit of normal.
10. Men and women of reproductive potential must agree to follow accepted birth control methods (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
11. Negative Beta HCG test within 30 days in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization). Pregnancy testing is not required for post-menopausal or surgically sterilized women.

Exclusion Criteria:

1. Patient with active CNS involvement with lymphoid malignancy.
2. Known infection with HIV, HTLV-I, Hepatitis B, or Hepatitis C.
3. Patients with other malignancies diagnosed within 2 years prior to study registration. Skin squamous or basal cell carcinoma are exceptions.
4. Active bacterial, viral or fungal infections.
5. History of stroke within 6 months prior to study registration.
6. A prior allogeneic stem cell transplant.
7. Patient has received other investigational drugs within 3 weeks before study registration.
8. Presence of circulating malignant lymphoid cells or bone marrow with lymphoma that constituted more than 25% of the cellular elements.
9. Serious nonmalignant or malignant disease or psychiatric illness, which, in the opinion of the investigator would compromise protocol objectives or interfere with participation.
10. Patients who are breast-feeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issa F. Khouri, MD,BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Yttrium-90 Ibritumomab + Chemo: Day -22 and -14, Rituximab 250 mg/m2 preceding In Ibritumomab and ibritumomab tiuxetan administration, respectively. Day -22, -21 to -16, Imaging, repeated 3-6 hours later (including Single Photon Emission-Computed Tomography/Computed Tomography (SPECT/CT) scan of the abdomen). Day -14,ibritumomab tiuxetan administration. Day -5, -4 and -3, Fludarabine and Bendamustine following Stem Cell Transplant (SCT) and CT. Fludarabine 30 mg/m2 intravenously followed by Bendamustine 130 mg/m2 intravenously. All patients receive Graft Versus Host Disease (GvHD) prophylaxis, infections disease prophylaxis, growth factors, blood and platelet transfusion and other supportive treatment.
Period: Overall Study
Arm/Group | Yttrium-90 Ibritumomab + Chemo
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Yttrium-90 Ibritumomab + Chemo
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Treatment-Related Mortality (TRM)
Description: Number of participants without treatment related mortality at day 100.
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Yttrium-90 Ibritumomab + Chemo
Number analyzed (Participants) | 20
Participants | 18

2. Secondary Outcome: Overall Survival (OS)
Description: Percentage of participants alive at 3 years.
Time Frame: From date of treatment to date of relapse or death, up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Yttrium-90 Ibritumomab + Chemo
Number analyzed (Participants) | 20
Participants | 14

ADVERSE EVENTS:
Time Frame: up to 3 years
Arm/Group | Yttrium-90 Ibritumomab + Chemo
All-Cause Mortality (participants affected / at risk) | 6/20
Serious Adverse Events (participants affected / at risk) | 12/20
Other Adverse Events (participants affected / at risk) | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Yttrium-90 Ibritumomab + Chemo (N=20)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Sepsis (Infections and infestations) | 1
Infections and Infestations (Infections and infestations) | 8
Thromboembolic (Vascular disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 8
Acute kidney injury (Renal and urinary disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Blood bilirubin increased (Investigations) | 1
Upper Respiratory Infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Yttrium-90 Ibritumomab + Chemo (N=20)
Nausea (Gastrointestinal disorders) | 17
Hypertension (Vascular disorders) | 4
Creatinine increased (Investigations) | 2
Fever (Infections and infestations) | 8
Diarrhea (Gastrointestinal disorders) | 6
Headache (Nervous system disorders) | 3
Infection (Infections and infestations) | 2
Thromboembolic (Vascular disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1
Weight gain (Investigations) | 4
Mucositis oral (Gastrointestinal disorders) | 7
Blood bilirubin increased (Investigations) | 1
Eye disorder (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT01490723/Prot_SAP_000.pdf